CLINICAL TRIAL: NCT00242073
Title: The Potential Use of BOLD MRI as a Noninvasive Measure of Tumor Hypoxia in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 02-0563-C
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Procedure: MRI Prostate

SUMMARY:
Hypoxia (low oxygen level) is know to be present in many tumors and may strongly influence the success of treatment and the progression of disease in prostate cancer. The method used to measure tumor oxygen levels in prostate cancer is to place a needle in the prostate itself through the rectum. Blood oxygen level dependent imaging (BOLD MRI) is a special MRI technique that allows indirect assessment of oxygen levels in blood. This technique is non-invasive, involving no needles. BOLD has not been applied in humans in prostate cancer. The purpose of this study is to develop a MRI-BOLD technique that allows us to non-invasively measure changes related to tumor hypoxia in prostate cancer. This technique may provide information that will be an independent predictor of patient survival, tumor recurrence and likelihood of treatment response in prostate cancer

DETAILED DESCRIPTION:
Hypoxia (low oxygen level) is know to be present in many tumors and may strongly influence the success of treatment and the progression of disease in prostate cancer. The method used to measure tumor oxygen levels in prostate cancer is to place a needle in the prostate itself through the rectum. Blood oxygen level dependent imaging (BOLD MRI) is a special MRI technique that allows indirect assessment of oxygen levels in blood. This technique is non-invasive, involving no needles. BOLD has not been applied in humans in prostate cancer. The purpose of this study is to develop a MRI-BOLD technique that allows us to non-invasively measure changes related to tumor hypoxia in prostate cancer. This technique may provide information that will be an independent predictor of patient survival, tumor recurrence and likelihood of treatment response in prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* prostate cancer

Exclusion Criteria:

* contraindication to MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masoom Haider, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada